CLINICAL TRIAL: NCT06611046
Title: Perfil De MicroRNA Como Biomarcador De Daño Hepático En Diferentes Tipos De Donantes De Hígado (MicroRNA Profile As a Biomarker of Liver Damage in Different Types of Liver Donors).
Brief Title: MicroRNA Profile As a Biomarker of Liver Damage in Different Types of Liver Donors.
Status: Completed | Type: Observational
Sponsor: Mar Dalmau (Other)
Collaborators: Vall Hebron Insitut Recerca (Network)
Responsible Party: Sponsor-Investigator, Mar Dalmau, Specialist in General Surgery and Digestive System, Hospital Vall d'Hebron
Organization: Hospital Vall d'Hebron (Other)
Other Study IDs: PR(AG)46/2019
Record Dates: First submitted 2024-09-19; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: MicroRNA Profile; Liver Transplant; Organ Donor
Keywords: microRNA; Liver donors; Liver transplant; heparinase

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — * Serum extracted from blood samples
  * Liver biopsies
  * Preservation solution fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Death brain donors (DBD): Liver grafts from brain death donors suffer systemic haemodynamic, inflammatory and endocrine changes during donor maintenance due to brain-stem activity cessation.
  Interventions: Other: organ donor
- Donors after circulatory death (DCD): Circulatory death donors do not suffer the physiologic features from brain death, almost mirroring a living donation. However, after withdrawal of life-sustaining measures these grafts suffer injury from severe ischemia.
  Interventions: Other: organ donor
- Discarded DBD (dDBD): Liver grafts from brain death donors that were unusable due to moderate to severe steatosis. Fatty livers are vulnerable to preservation injury resulting in a higher rate of primary non-function, early allograft dysfunction and post-transplant vascular and biliary complications
  Interventions: Other: organ donor
- Control group: Serum samples from healthy patients who underwent elective cholecystectomy due to symptomatic gallstones were collected before incision. The patients included shared similar characteristics according to the centre living liver donor policy: 18 to 60-year-old, normal liver function and no steatosis in ultrasound.
  Interventions: Other: organ donor

INTERVENTIONS:
Other: organ donor — Observational study with sample collection of serum, liver tissue and perfusate fluid from liver donors. No specific interventions were done to the donors as part of the study. The samples were analyzed for specific microNA expression by RT-qPCR.
  *Control group: only serum samples were collected from this group.

SUMMARY:
The goal of this observational study is to analyze the expression of liver-derived miRNAs in different types of liver donors to gain in depth knowledge about distinctive physiologic features within donors and find potential biomarkers for graft quality assessment. The main questions it aims to answer are:

Is there a distinctive miRNA profile between donors after brain-stem death and donors after circulatory death?

Is heparinase I treatment necessary to overcome miRNA quantification interference in heparinized liver donor samples ?

Researchers will compare miRNA expression in donors after brain-stem death and donors after circulatory death with I) a subgroup of donors with unusable grafts due to significant steatosis, 2) and with a subgroup of healthy controls undergoing elective cholecystectomy to set the reference miRNA profiles in extreme conditions.

DETAILED DESCRIPTION:
Between October 2019 and May 2021, perfusates, liver biopsies and serum samples were collected prospectively from adult deceased organ donors in Vall d'Hebron University Hospital, Barcelona, Spain.

Samples from adult human brain death donors (n=10) and donors after circulatory death (n=10) were analyzed for the presence of miR-122, miR-148, miR-155, miR-22, miR-222 and ratio miR122/miR222, target biomarkers of liver injury selected from the literature.

To set the reference miRNA profiles, a subgroup of donors with unusable grafts due to significant steatosis (n=3) were analyzed.

Donors for re-transplantation, pediatric, and split were excluded to avoid biopsy-related injury.

As there were no living donor inclusions in the study period, serum specimens from a subgroup of healthy controls undergoing elective cholecystectomy (n=7) were analyzed.

This study is part of a PhD thesis and data collection was done by the main investigator based in organ donor availability in one tertiary hospital centre in Barcelona, Spain. Based on resource limitation constraints, the sample size was limited to the consecutive samples obtained in a 2-year period.

Written informed consent was obtained from patients and relatives of donors included in the study. Samples and data from patients were provided by the Vall d'Hebron University Hospital Biobank (PT20/00107), integrated in the Spanish National Biobanks Network, and they were processed following standard operating procedures. The study protocol was approved by the medical ethics committee of the Vall d'Hebron University Hospital [PR(AG)46/2019] and conforms to the principles outlined in the Declaration of Helsinki.

Statistical analysis:

To optimize the quality of data, readings with extreme Ct values (Ct less than 11 or Ct greater than 39) were discarded. The mean of the Cts and the standard deviation for each of the miRNAs in the different samples analyzed (technical triplicates) were calculated. To improve the quality of the data analyzed, in triplicates with high standard deviation (Ct SD greater than 0.3), the Ct value furthest from the mean was eliminated, leaving a total of at least two values per miRNA per sample. Likewise, for each miRNA, samples with less than two valid replicates were excluded. To correct for potential RNA input or RT efficiency biases, Ct values were normalized using the average Ct of endogenous references (miR-103a, miR-191, miR-30c, miR-16 and let7a). miRNA relative quantification (RQ) levels were analyzed using the Livak et al. method 2^(-ΔΔCt), calculated as follows ΔCt (miRNA Ct target - averaged endogenous control Ct) and the difference (ΔΔCt) between comparison groups (ΔCt comparison - ΔCt reference sample. Group comparisons were performed using T-test or U-Mann Whitney (non-parametric) for continuous data and Fisher test for qualitative. P-values less than 0.05 were considered significant.

Methodology substudy:

A subgroup of adult human brain death donors (n=4) and donors after circulatory death (n=4) were analyzed for the presence of miR-122 and miR-148. Heparin is known to have an inhibiting effect in RNA qPCR analysis and liver donor samples are prone to have heparin traces, as it's used to avoid thrombus formation during organ procurement. Heparinase-I has been used in the literature to overcome the heparin inhibiting effect.

In this substudy, the samples were treated with 0 IU, 6 IU or 12 IU of heparinase-I to evaluate the counteracting effect of heparinase I on miRNA detection levels by RT-qPCR.

ELIGIBILITY:
I) Main donor groups (DBD and DCD):

Inclusion Criteria:

* Adult deceased liver donors

Exclusion Criteria:

* Pediatric donors (less than18 year-old)
* Donors for re-transplantation cases
* Donors who underwent split or partition liver technique to obtain two small grafts for two recipients (adult and pediatric).

II) Discarded DBD grafts:

Inclusion Criteria:

- Unusable grafts for transplantation due to moderate (30% to 60%) or severe (more than 60%) steatosis in liver biopsies.

Exclusion Criteria:

* Unusable grafts discarded for other reasons.
* Pediatric donors (less than18 year-old)
* Donors for re-transplantation cases
* Donors who underwent split or partition liver technique to obtain two small grafts for two recipients (adult and pediatric).

III) Control group:

Inclusion criteria:

- Same inclusion criteria as the living liver donor program in our center: 18 to 60 years old, normal liver function, ultrasound without signs of liver disease and steatosis less than 30%.

Exclusion criteria:

- Patients with preoperative deranged liver function tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fourteen combined perfusates, liver biopsies and serum samples were collected prospectively from brain death donors (DBD, n=14) and donors after circulatory death (DCD, n=14).
  Three combined perfusates, liver biopsies and serum samples were collected prospectively from brain death donors discarded for transplantation due to significant steatosis (DBDd, n=3).
  Seven serum samples were collected prospectively from healthy controls undergoing elective cholecystectomy (Control, n=7).
  Single centre study with samples collected at Vall d'Hebron University Hospital, Spain, between October 2019 and May 2021.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
miRNA expression profile in different types of liver donors. | Data collection from regional donors in a period of two years based on donor availability and main investigator (data collector) availability. The samples were collected during organ procurement which entails over 4 to 6 hours in each donor.
  Compare the miRNA expression profile (miR-122 and miR-148a, miR-222, miR-22 and miR-155) from death brain donors and circulatory death donors in liver biopsies, serum and perfusion solution

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Charco, MD, PhD, Study Director — Chief of HPB surgery and Transplant Department in Vall d Hebron University Hospital; Concepción Gómez-Gavara, MD, PhD, Study Director — HPB surgery and Liver Transplant consultant in Vall d Hebron University Hospital
Locations (1):
- Vall d Hebron University Hospital, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dalmau M, Charco R, Bilbao I, Dopazo C, Caralt M, Molino JA, Gomez-Gavara C. Heparinase I treatment to overcome RNA quantification interference in heparinized liver donor samples: One size fits all? PLoS One. 2025 May 12;20(5):e0322899. doi: 10.1371/journal.pone.0322899. eCollection 2025. PMID 40354476